CLINICAL TRIAL: NCT07342907
Title: Effectiveness of Internal Family Systems Therapy in Improving Mental Health in Individuals With Borderline Personality Disorder
Brief Title: Internal Family Systems Therapy for Borderline Personality Disorder
Acronym: IFS for BPD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Waypoint Centre for Mental Health Care (Other)
Responsible Party: Principal Investigator, Barna Konkoly-Thege, Research Psychologist, Waypoint Centre for Mental Health Care
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IFS for BPD
Record Dates: First submitted 2026-01-06; First posted 2026-01-15 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Borderline Personality Disorder (BPD)
Keywords: borderline personality disorder; psychotherapy; effectiveness; internal family systems therapy
MeSH Terms: conditions — Borderline Personality Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention recipients (Experimental): Participants will engage in internal family systems therapy in the individual format. This form of psychotherapy conceptualizes the mind as a system of subpersonalities ('parts') organized around a compassionate, stable core Self. The approach promotes internal harmony through increasing awareness, acceptance, and cooperation among these parts and the Self. Participants will receive weekly, up to 50, one-hour IFS therapy sessions in the private mental health care setting over approximately 12 to 15 months. Treatment will be delivered by two licensed mental health professionals trained in the IFS model. Participants will pay a significantly subsidized session fee to reduce financial burden of participation in the intervention.
  Interventions: Behavioral: Internal family systems therapy

INTERVENTIONS:
Behavioral: Internal family systems therapy — The internal family systems model was developed by Richard C. Schwartz in the 1980s. This psychotherapy is based on the assumption that the human mind is naturally multiple and consists of interacting sub-personalities ("parts"), including protective and vulnerable parts, shaped by development and adversity. All parts are assumed to have positive intentions, even when their effects are maladaptive; therapy therefore aims to transform rather than eliminate them. Internal family systems therapy further posits the existence of a core Self in every person, characterized by qualities such as compassion, clarity, and calm, which is inherently intact in each individual and capable of leading the internal system. Therapeutic change involves increasing the leadership skills of the core Self, building trusting relationships among parts and the core Self, and unburdening vulnerable parts so they can assume more adaptive roles, supporting improved emotion regulation and well-being.
  Other Names: IFS

SUMMARY:
Borderline Personality Disorder (BPD) involves intense emotional ups and downs, unstable relationships, impulsivity, and a poor sense of self. These challenges often lead to addiction, self-harm, and frequent use of healthcare services. While certain treatments already in practice - such as dialectical behavior therapy - can help, they don't work for everyone or address all aspects of the disorder. This study plans to explore internal family systems (IFS) therapy, a method that views the mind as made up of different "parts" - each with its own thoughts and feelings. IFS helps people build understanding and compassion toward these parts and connect with a calmer, more centered "Self." This may be especially useful for those with BPD, who often feel fragmented and extremely critical of themselves and others. This will be the first study to examine internal family systems therapy for BPD. The participants (15 in total) will receive up to 50 individual sessions over 15 months. Changes in symptoms and overall mental health will be measured at four points during the study. People with lived experience of BPD will help shape the research to ensure it is relevant, respectful, and useful for others facing similar challenges.

DETAILED DESCRIPTION:
Brief background and rationale: Borderline personality disorder (BPD) is a chronic and disabling psychiatric condition marked by pervasive affective instability, identity disturbance, interpersonal dysfunction, and impulsivity. It affects approximately 1-2% of the general population and up to 20% of psychiatric populations, contributing substantially to healthcare utilization, suicide risk, and long-term disability. Existing evidence-based psychotherapies for this condition, such as dialectical behavior therapy, mentalization-based therapy, or schema therapy show significant benefits but these are modest and these interventions are quite resource-intensive. There remains a need for additional, theoretically grounded treatments that target core pathomechanisms of BPD-particularly emotion dysregulation, shame, and self-fragmentation.

Objectives: The primary objective of this pilot study is to assess preliminary effectiveness of internal family systems (IFS) therapy in reducing BPD symptom severity from baseline to post-treatment. Secondary objectives are to evaluate changes in emotion dysregulation, shame, self-compassion, interpersonal functioning, depression, anxiety, addictive behaviors and overall well-being; as well as to assess feasibility (recruitment, retention, adherence), acceptability, and safety. It is hypothesized that participants will demonstrate at least small-to-moderate improvements in BPD symptom severity, with congruent changes across secondary outcomes. Although clinical interest in IFS has grown exponentially in the past decades, empirical evaluation remains limited, and no studies to date have specifically examined its use in any personality disorder. Given the strong theoretical fit between IFS principles and BPD phenomenology, a structured pilot investigation is warranted to establish feasibility, safety, and preliminary effectiveness prior to larger controlled trials.

Study design: The study will use a single-group, repeated-measures design with assessments at baseline, 4 months, 8 months, and post-intervention (12-15 months). A target sample of fifteen adults will be recruited. Inclusion criteria are age 18 or older, sufficient English proficiency for participation, and a formal BPD diagnosis confirmed by a referring clinician. Exclusion criteria include active psychosis or mania, cognitive impairment, inadequate English comprehension, or participation in another form of psychotherapy during the study period.

Intervention: Internal family systems therapy, developed by Richard Schwartz, is an integrative psychotherapy that conceptualizes the mind as a system of subpersonalities ('parts') organized around a compassionate, stable core Self. The approach promotes internal harmony through increasing awareness, acceptance, and cooperation among these parts and the Self. Participants will receive weekly, one-hour IFS therapy sessions in the private mental health care setting over approximately 12 to 15 months. Treatment will be delivered by two licensed mental health professionals trained in the IFS model. Participants will pay a significantly subsidized session fee to reduce financial burden of participation in the intervention.

Outcomes: The primary outcome is BPD symptom severity measured by the Borderline Symptom List-23 and its supplement. Secondary outcomes include validated measures of emotion dysregulation (DERS-18), shame and guilt (GSQ-8), self-compassion (SCS-SF), interpersonal functioning (EXIS.pers), depression (PHQ-9), anxiety (GAD-7), addictive behaviors (SSBA-G), and well-being (WHO-5). Feasibility and acceptability will be evaluated through attendance, retention, and brief structured questionnaires.

Data collection and analysis: Data will be collected electronically via REDCap, using unique participant IDs and secure storage protocols. Analyses will include paired t-tests for pre-post differences and linear mixed-effects models for repeated measures across all four time points. Effect sizes will be prioritized over probability values when interpreting the results considering relatively low anticipated statistical power.

Timeline: The study begins in early 2026 following ethics approval, with recruitment and intervention delivery extending through the end of 2027. Data analysis, manuscript preparation, and dissemination are planned for 2028.

ELIGIBILITY:
Inclusion Criteria:

* Resident of Ontario, Canada;
* Sufficient fluency in English to provide informed consent, participate in therapy sessions, and complete self-reported assessments;
* Diagnosis of borderline personality disorder confirmed by a healthcare professional authorized to establish such a diagnosis in Ontario;
* Willingness and ability (including financial means) to participate in the 50-session, 12-15-month intervention and the study assessments;
* Capacity and willingness to provide written informed consent.

Exclusion Criteria:

* Current manic or psychotic symptoms regardless of diagnosis;
* Substance dependence severe enough to interfere with meaningful level of engagement in the study intervention.
* Cognitive impairment or neurological disorders that would preclude informed consent or meaningful participation in the study intervention.
* Concurrent participation in any another form of psychotherapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Severity of borderline personality disorder symptomatology - disorder-specific mental distress | Change in scores between baseline and intervention end (approx. 12-15 months)
  This first indicator of the primary outcome will be assessed by the Borderline Symptom List (BSL-23, Bohus et al., 2009). This self-report measure consists of items that 1) are based on DSM diagnostic criteria as well as expert opinions and expert-by-experience input; and 2) displayed a high level of sensitivity to change and ability to discriminate individuals with versus without borderline personality disorder. Scale items cover areas such as affective instability, emotional pain, identity disturbance, interpersonal sensitivity, cognitive-perceptual distress, impulsivity-related subjective distress, and suicidal ideation. Total scores range from 0 to 92 with higher scores indicating greater severity of borderline personality disorder symptoms.
Severity of borderline personality disorder symptomatology - dysfunctional behaviors | Change in scores between baseline and intervention end (approx. 12-15 months)
  This second indicator of the primary outcome will be assessed by the supplementary scale of the Borderline Symptom List (BSL). This 11-item scale (BSL-Supplement; Bohus et al., 2007) assesses the extent of dysfunctional behaviours associated with borderline personality disorder such as self-injurious behaviour, suicidality, binge and purge behaviours, impulsivity, hostile outbursts, and sexual promiscuity. Total scores range from 0 to 44 with higher scores reflecting greater frequency or severity of borderline-related behaviors.

SECONDARY OUTCOMES:
Emotion dysregulation | Change in scores between baseline and intervention end (approx. 12-15 months)
  Emotion dysregulation will be assessed using the abbreviated, 18-item version of the Difficulties in Emotion Regulation Scale (DERS-18). The DERS-18 is a self-report measure that captures key dimensions of emotion dysregulation, including lack of emotional clarity, nonacceptance of emotional responses, difficulties engaging in goal-directed behavior, impulse control difficulties, and limited access to effective regulation strategies. Total scores range from 18 to 90, with higher scores indicating greater emotion dysregulation. Despite its brevity, the DERS-18 demonstrates strong psychometric properties and retains coverage of the core domains assessed by the original full-length version (Gratz & Roemer, 2004).
Addictive behaviors | Change in scores between baseline and intervention end (approx. 12-15 months)
  Addictive behaviours will be assessed using the Generalized Version of the Screener for Substance and Behavioural Addictions (SSBA-G). The SSBA-G is an 8-item, transdiagnostic self-report tool that screens for engagement in and perceived problematic use of a broad range of substances and behaviours (Konkolÿ Thege et al., 2023). Total scores range from 8 to 56, with higher scores indicating more severe addiction-related problems. This tool was selected over disorder- or substance-specific instruments due to its comprehensive scope, brevity, and ability to capture cross-addiction tendencies often observed in the target population.
Interpersonal functioning | Change in scores between baseline and intervention end (approx. 12-15 months)
  Interpersonal functioning will be assessed by the Experience in Personal Social Systems Questionnaire (Hunger et al., 2017). This 12-item scale covers four dimensions in relation to 1) belonging (a sense of being part of a social system); 2) autonomy (ability to demark boundaries based on the belief that the renegotiation of roles, rights, and responsibilities is possible); 3) accord (acceptance of one's social system the way as it is); and 4) confidence (trust in the individual's and their social system's ability to cope with emerging difficulties). Total scores range from 12 to 72, with higher scores indicating better interpersonal functioning. This scale demonstrated good psychometric properties and sensitivity to change in intervention studies. This measure was chosen due to its positive approach to interpersonal functioning (instead of a focus on pathology) and brevity compared to other measures assessing interpersonal functioning.
Shame and guilt | Change in scores between baseline and intervention end (approx. 12-15 months)
  The Guilt and Shame Questionnaire (GSQ-8) is a brief, validated self-report instrument designed to assess the frequency of guilt and shame experiences in the past month (Hoppen et al., 2022). The scale consists of 8 items-four assessing guilt and four assessing shame-rated on a Likert scale. It has demonstrated good internal consistency and a stable two-factor structure across clinical and non-clinical samples. Total scores range from 0 to 32, with higher scores indicating greater levels of guilt and shame. The GSQ-8 is sensitive to changes in self-conscious emotions and provides a concise, practical tool for repeated use in clinical research.
Self-compassion | Change in scores between baseline and intervention end (approx. 12-15 months)
  The Self-Compassion Scale - Short Form (SCS-SF) is a 12-item self-report measure that assesses six key components of self-compassion: self-kindness, self-judgment, common humanity, isolation, mindfulness, and over-identification (Raes et al., 2011). The recommended indicator for this scale is the mean of all items, which score ranges from 1 to 5, with higher scores indicating greater self-compassion. The SCS-SF has demonstrated strong psychometric properties, including good internal consistency and high correlation with the original long-form version.
Anxiety | Change in scores between baseline and intervention end (approx. 12-15 months)
  The Generalized Anxiety Disorder-7 (GAD-7) is a 7-item self-report questionnaire that measures the severity of generalized anxiety symptoms over the past two weeks (Spitzer et al., 2006). Total scores range from 0 to 21, with higher scores indicating more severe anxiety symptoms. The GAD-7 is brief and has been extensively validated in both general and clinical populations. It has demonstrated good internal consistency, construct validity, and responsiveness to treatment, making it an appropriate tool for evaluating anxiety outcomes in BPD intervention studies.
Depression | Change in scores between baseline and intervention end (approx. 12-15 months)
  The Patient Health Questionnaire-9 (PHQ-9) is a widely used, brief self-report measure that assesses the severity of depressive symptoms over the past two weeks (Kroenke, Spitzer, & Williams, 2001). It consists of nine items corresponding to DSM-5 diagnostic criteria for major depressive disorder. Total scores range from 0 to 27, with higher scores indicating more severe depressive symptoms. The PHQ-9 is well-validated across clinical populations, including those with comorbid personality disorders, and demonstrates strong reliability, sensitivity to change, and diagnostic utility.
General psychological well-being | Change in scores between baseline and intervention end (approx. 12-15 months)
  The WHO-5 Well-Being Index is a widely used, validated self-report measure that assesses current mental well-being (World Health Organization, 2024). It consists of five positively worded items related to mood, vitality, and general interest in life. Raw scores range from 0 to 25 (0-100 when transformed as recommended by the developer), with higher scores indicating greater subjective well-being. The WHO-5 is brief, easy to administer, and sensitive to change, making it suitable for both clinical and research settings.

OTHER OUTCOMES:
Intervention feasibility | Intervention end only (approx. 12-15 months)
  It will be captured how many participants initiated versus completed the intervention (defined as attending ≥70% of the 50 therapy sessions offered). Higher proportion of completers indicates better feasibility.
Intervention tolerability | Intervention end only (approx. 12-15 months)
  Rating [from 0 (no distress) to 10 (extreme distress)] in relation to the question: "How difficult or distressing did you find participating in the therapy you received as part of this study?" Higher scores are indicative of worse tolerability.
Intervention satisfaction | Intervention end only (approx. 12-15 months)
  Rating [from 0 (not at all satisfied) to 10 (extremely satisfied)] in relation to the question: "Overall, how satisfied are you with the therapy you received as part of this study?" Higher scores are indicative of greater service user satisfaction.
Intervention relevance | Intervention end only (approx. 12-15 months)
  Rating [from 0 (not at all relevant) to 10 (extremely relevant)] in relation to the question: "What do you think, how relevant this specific form of therapy (focus on internal parts and their relationship to each other and the Self) was to your particular mental health condition?" Higher scores are indicative of greater intervention relevance for the target population.
Perceived intervention effectiveness | Intervention end only (approx. 12-15 months)
  Rating [from -5 (worsened significantly) to 5 (improved significantly)] in relation to the question: "What is your overall impression, how your mental health has changed (if at all) as a result of the therapy you received as part of this study?" Higher scores are indicative of greater perceived intervention effectiveness.

CONTACTS AND LOCATIONS:
Overall Officials: Barna Konkoly-Thege, PhD, Principal Investigator — Waypoint Centre for Mental Health Care
Locations (1):
- Provincewide across Ontario (intervention can be delivered virtually), Tiny, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
A public repository dataset will be created from the anonymized data of those participants only who provided explicit consent during the informed consent process to allow their data to be stored in a data repository for secondary analyses. This dataset will be uploaded to a controlled-access repository (University of Toronto Dataverse within the Borealis network).
Supporting Information: Study Protocol, ICF
Time Frame: The data set will be available upon study completion, permanently.